CLINICAL TRIAL: NCT02513459
Title: An Open Label, Single Group, Long Term Safety Extension Trial of BI 655066/ABBV-066 (Risankizumab), in Patients With Moderately to Severely Active Crohn's Disease
Brief Title: A Long Term Extension Trial of BI 655066/ABBV-066 (Risankizumab), in Patients With Moderately to Severely Active Crohn's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M15-989; 2015-001834-15 (EudraCT Number); 1311.2 (Other Grant/Funding Number: Boehringer Ingelhem)
Expanded Access: NCT03914261 (No longer available)
Record Dates: First submitted 2015-07-30; First posted 2015-07-31 (Estimated); Results first posted 2020-04-24 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Crohn Disease
Keywords: ABBV-066; BI 655066; Risankizumab
MeSH Terms: conditions — Crohn Disease | interventions — risankizumab

STUDY DESIGN:
Intervention Model Description: Participants with clinical response or remission at the end of Study NCT02031276 (Boehringer Ingelheim trial 1311.6/AbbVie M15-993) or at screening for this study were rolled over directly into this study and received maintenance therapy of risankizumab 180 mg administered subcutaneously (SC) every 8 weeks (q8w) from Visit 2 through the end of trial (EOT) visit. Participants who lost response or remission between the completion of Study NCT02031276 and enrollment in this study received open-label intravenous (IV) re-induction treatment with risankizumab consisting of 3 infusions of 600 mg IV every 4 weeks (q4w), after which eligibility was assessed if clinical response was re-gained. If clinical response or remission was achieved, participants continued with maintenance treatment of risankizumab 180 mg SC q8w beginning at Visit 5.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Risankizumab (Experimental): Maintenance treatment with risankizumab 180 mg administered subcutaneously (SC) every 8 weeks (q8w) from Visit 2 through the end of trial (EOT) visit. Participants who re-gained their clinical response following the re-induction treatment could continue with maintenance treatment beginning at Visit 5.
  Interventions: Drug: Risankizumab 600 mg IV; Drug: Risankizumab 180 mg SC

INTERVENTIONS:
Drug: Risankizumab 600 mg IV — Re-induction treatment; 3 infusions every 4 weeks, after which eligibility was assessed if clinical response was re-gained
  Other Names: BI 655066; ABBV-066
Drug: Risankizumab 180 mg SC — Maintenance treatment every 8 weeks (q8w) from Visit 2 through the end of trial (EOT) visit. Participants who re-gained their clinical response following the re-induction treatment could continue with maintenance treatment beginning at Visit 5.
  Other Names: BI 655066; ABBV-066

SUMMARY:
The primary objective of the study was to investigate long-term safety of risankizumab (BI 655066/ABBV-066) in participants with moderately to severely active Crohn's disease who showed a clinical response or remission on previous treatment with risankizumab in Study NCT02031276 (BI trial 1311.6/ AbbVie M15-993) and were now receiving long-term treatment. Additional objectives of this study were to further investigate long-term efficacy, tolerability, pharmacokinetics, pharmacodynamics and immunogenicity of risankizumab.

DETAILED DESCRIPTION:
This was a single group, open-label long-term extension study that assessed the long-term safety, efficacy, and pharmacokinetics of risankizumab in participants with moderately to severely active Crohn's disease. This study was terminated early by AbbVie to enable participants who completed the study to rollover into Study NCT03105102 (AbbVie M16-000 Sub-Study 3 [Phase 3 OLE study]) for further OLE treatment within the Phase 3 program, which allows for risankizumab dose escalation if needed.

ELIGIBILITY:
Inclusion Criteria:

* Participants with Crohn's disease, who had successfully completed the preceding trial NCT02031276 (Boehringer Ingelheim trial 1311.6/AbbVie M15-993). Successful treatment is defined as:

  1. Completion of period 2 in 1311.6 with a clinical response (drop in Crohn's Disease Activity Index (CDAI) from baseline by ≥100) but no remission (CDAI < 150) at Visit E1; or
  2. Completion of period 3 in 1311.6 with a clinical response (drop in CDAI from baseline by ≥100) and/or remission (CDAI < 150) at Visit E5; or
  3. Completion of period 2 or 3 in 1311.6 per protocol with a clinical response or remission before initiation of 1311.20 can roll-over either directly if that response/remission is maintained or through an open-label i.v. re-induction phase if they have lost their previous response/remission.
* Female participants:

  1. Women of childbearing potential (not surgically sterilized and between menarche and 1 year postmenopause), that, if sexually active agree to use one of the appropriate medically accepted methods of birth control in addition to the consistent and correct use of a condom from date of screening until 20 weeks after last administration of study medication. Medically accepted methods of contraception are: ethinyl estradiol containing contraceptives, diaphragm with spermicide substance, and intrauterine device, or
  2. Surgically sterilized female participants with documentation of prior hysterectomy, tubal ligation or complete bilateral oophorectomy, or
  3. Postmenopausal women with postmenopausal is defined as permanent cessation >/=1 year of previously occurring menses, and
  4. Negative serum ß-Human Chorionic Gonadotrophin test at screening and urine pregnancy test prior to randomization.
* Male participants:

  1. Who are documented to be sterile, or
  2. Who consistently and correctly use effective method of contraception (i.e. condoms) during the study and 20 weeks after last administration of study medication.
* Be able to adhere to the study visit schedule and other protocol requirements.

Exclusion Criteria:

* Participants who were not compliant with key study procedures (colonoscopy, treatment compliance, endpoint assessment, contraception measures) in preceding trial 1311.6
* Participants who could not tolerate risankizumab (BI 655066/ ABBV-066) treatment for tolerability or safety reasons in the preceding trial
* Are pregnant, nursing, or planning pregnancy while enrolled in the study, or within 20 weeks after receiving the last dose of study medication.
* Participants must agree not to receive a live virus or bacterial or Bacille Calmette-Guérin vaccination during the study or up to 12 months after the last administration of study drug.
* Participants who have developed malignancy, or suspicion of active malignant disease during the preceding trial
* Are intending to participate in any other study using an investigational agent or procedure during participation in this study.
* Cannot adhere to the concomitant medication requirements

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2015-09-16 (Actual); Primary Completion 2019-06-19 (Actual); Study Completion 2019-06-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (28):
- United States (2):
  - MGG Group, Inc.Chevy Chase Clinical Research /ID# 155068, Chevy Chase, Maryland
  - Clin Res Inst of Michigan, LLC /ID# 155066, Chesterfield, Michigan
- Belgium (7):
  - Cliniques Universitaires Saint Luc /ID# 154985, Woluwe-Saint-Lambert, Brussels Capital
  - CHU de Liege /ID# 154988, Liège, Liege
  - Imelda Ziekenhuis /ID# 154984, Bonheiden
  - ULB Erasme /ID# 154987, Brussels
  - AZ Groeninge /ID# 154989, Kortrijk
  - UZ Leuven /ID# 154986, Leuven
  - AZ-Delta /ID# 154983, Roeselare
- McMaster University Med Cent /ID# 155019, Hamilton, Ontario, Canada
- Germany (2):
  - Universitaetsklinikum Erlangen /ID# 155039, Erlangen, Bavaria
  - Med Hochschule Hanover /ID# 155041, Hanover
- Netherlands (2):
  - Academisch Medisch Centrum /ID# 155058, Amsterdam, North Holland
  - Maastricht Universitair Medisch Centrum /ID# 155059, Maastricht
- Poland (2):
  - NZOZ Vivamed /ID# 155061, Warsaw
  - Lexmedica /Id# 155062, Wroclaw
- South Korea (4):
  - Yeungnam University Med Ctr /ID# 155056, Daegu, Daegu Gwang Yeogsi
  - Kangbuk Samsung Hospital /ID# 155054, Jongno-Gu, Seoul Teugbyeolsi
  - Severance Hospital /ID# 155055, Seoul, Seoul Teugbyeolsi
  - Asan Medical Center /ID# 155053, Seoul
- Spain (3):
  - Hospital Duran i Reynals /ID# 155063, L'Hospitalet de Llobregat, Barcelona
  - Hospital Clinic de Barcelona /ID# 155064, Barcelona
  - Hospital Univ de la Princesa /ID# 155065, Madrid
- United Kingdom (5):
  - Guy's and St Thomas' NHS Found /ID# 155046, London, London, City of
  - Addenbrookes Hospital /ID# 155047, Cambridge
  - St. James University Hospital /ID# 155050, Leeds
  - The Newcastle Upon Tyne Hospitals NHS Foundation Trust' /ID# 155049, Newcastle upon Tyne
  - John Radcliffe Hospital /ID# 155048, Oxford

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Data requests can be submitted at any time and the data will be accessible for 12 months, with possible extensions considered.
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information on the process, or to submit a request, visit the following link.
URL: https://www.abbvie.com/our-science/clinical-trials/clinical-trials-data-and-information-sharing/data-and-information-sharing-with-qualified-researchers.html

REFERENCES:
- [Derived] Ferrante M, Feagan BG, Panes J, Baert F, Louis E, Dewit O, Kaser A, Duan WR, Pang Y, Lee WJ, Gustafson D, Liao X, Wallace K, Kalabic J, D'Haens GR. Long-Term Safety and Efficacy of Risankizumab Treatment in Patients with Crohn's Disease: Results from the Phase 2 Open-Label Extension Study. J Crohns Colitis. 2021 Dec 18;15(12):2001-2010. doi: 10.1093/ecco-jcc/jjab093. PMID 34077509

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All enrolled participants
Groups:
- All Risankizumab: Participants who received at least one dose of risankizumab in the current study
Period: Overall Study
Arm/Group | All Risankizumab
Started | 65
Completed | 44
Not Completed | 21
Not completed — Adverse Event | 7
Not completed — Withdrew consent | 5
Not completed — Loss of efficacy | 2
Not completed — Pregnancy | 2
Not completed — Subject decision | 2
Not completed — Lack of response | 1
Not completed — Reproductive plans | 1
Not completed — Surgery planned-- not done | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat population: all participants who received at least one dose of risankizumab in the current study
Arm/Group | All Risankizumab
Number analyzed (Participants) | 65
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.1 (12.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 29
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 10
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 55
  More than one race | 0
  Unknown or Not Reported | 0
Baseline Corticosteroid Use [Count of Participants; unit: Participants]
  Yes | 21
  No | 44
  Missing | 0
Tumor Necrosis Factor (TNF) Antagonist Exposure [Count of Participants; unit: Participants]
  Anti-TNF Experienced | 60
  Anti-TNF Naive | 5
  Missing | 0
Crohn's Disease Activity Index (CDAI) [Mean (Standard Deviation); unit: units on a scale] — The Crohn's Disease Activity Index (CDAI) is a composite instrument that includes participant symptoms evaluated over 7 days (abdominal pain, stool frequency and general well-being), as well as physical and laboratory findings. These items are scored individually, weighted, and do not contribute equally to the overall score. The CDAI is derived from summing up the weighted individual scores of eight items. CDAI approximately ranges from 0 to 600 with higher scores indicating more severe disease.
  units on a scale | 304.771 (77.9832)
High-sensitivity C-Reactive Protein (hs-CRP) [Mean (Standard Deviation); unit: mg/L] | 20.315 (23.1676)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: A treatment emergent adverse event was defined as an event that occurred or worsened on or after the first dose of study drug through 140 days after the last dose in the current study for participants not rolling over into M16-000 Sub-study 3 or until the first dose of study drug in NCT03105102. All treatment-emergent serious and nonserious adverse events were collected, whether elicited or spontaneously reported by the participant.
Time Frame: From the time of study drug administration until 140 days after the last dose of study drug in the current study or until the first dose of study drug in NCT03105102 (AbbVie M16-000 Sub-study 3), up to 4 years for participants who rolled-over
Population: All participants who received at least one dose of risankizumab in the current study
Measure: Count of Participants; unit: Participants
Arm/Group | Risankizumab 600 mg IV | Risankizumab 180 mg SC | All Risankizumab
Number analyzed (Participants) | 4 | 65 | 65
Participants | 2 | 60 | 60

2. Secondary Outcome: Percentage of Participants Achieving Crohn's Disease Activity Index (CDAI) Clinical Remission by Visit
Description: The Crohn's Disease Activity Index (CDAI) is a composite instrument that includes participant symptoms evaluated over 7 days (abdominal pain, stool frequency and general well-being), as well as physical and laboratory findings. These items are scored individually, weighted, and do not contribute equally to the overall score. The CDAI is derived from summing up the weighted individual scores of eight items. CDAI approximately ranges from 0 to 600 with higher scores indicating more severe disease. Clinical remission is defined as CDAI score < 150.
Time Frame: Weeks 0, 4, 8, 16, 24, 32, 40, 48, 56, 64, 72, 80, 88, 96, 104, 112, 120, 128, 136, 144, 152, 160, 168, 176, and 184
Population: Observed case (OC) analysis was performed on the intent-to-treat (ITT) analysis sets. The ITT set for IV consisted of all participants who received at least one dose of risankizumab IV in the current study, and the ITT set for SC consisted of all participants who received at least one dose of risankizumab SC in the current study.
Measure: Number; unit: percentage of participants
Arm/Group | Risankizumab 600 mg IV | Risankizumab 180 mg SC
Number analyzed (Participants) | 4 | 65
percentage of participants
  Week 0 | 25.00 | 72.31
  Week 4: number analyzed (Participants) | 4 | 0
  Week 4 | 25.00 |
  Week 8 | 25.00 | 73.85
  Week 16: number analyzed (Participants) | 0 | 64
  Week 16 |  | 71.88
  Week 24: number analyzed (Participants) | 0 | 63
  Week 24 |  | 74.60
  Week 32: number analyzed (Participants) | 0 | 61
  Week 32 |  | 78.69
  Week 40: number analyzed (Participants) | 0 | 60
  Week 40 |  | 81.67
  Week 48: number analyzed (Participants) | 0 | 58
  Week 48 |  | 79.31
  Week 56: number analyzed (Participants) | 0 | 57
  Week 56 |  | 80.70
  Week 64: number analyzed (Participants) | 0 | 55
  Week 64 |  | 87.27
  Week 72: number analyzed (Participants) | 0 | 54
  Week 72 |  | 83.33
  Week 80: number analyzed (Participants) | 0 | 53
  Week 80 |  | 79.25
  Week 88: number analyzed (Participants) | 0 | 51
  Week 88 |  | 78.43
  Week 96: number analyzed (Participants) | 0 | 52
  Week 96 |  | 84.62
  Week 104: number analyzed (Participants) | 0 | 49
  Week 104 |  | 85.71
  Week 112: number analyzed (Participants) | 0 | 48
  Week 112 |  | 87.50
  Week 120: number analyzed (Participants) | 0 | 48
  Week 120 |  | 83.33
  Week 128: number analyzed (Participants) | 0 | 46
  Week 128 |  | 86.96
  Week 136: number analyzed (Participants) | 0 | 39
  Week 136 |  | 76.92
  Week 144: number analyzed (Participants) | 0 | 37
  Week 144 |  | 78.38
  Week 152: number analyzed (Participants) | 0 | 30
  Week 152 |  | 76.67
  Week 160: number analyzed (Participants) | 0 | 23
  Week 160 |  | 78.26
  Week 168: number analyzed (Participants) | 0 | 17
  Week 168 |  | 70.59
  Week 176: number analyzed (Participants) | 0 | 10
  Week 176 |  | 60.00
  Week 184: number analyzed (Participants) | 0 | 5
  Week 184 |  | 40.00

3. Secondary Outcome: Percentage of Participants Achieving Crohn's Disease Activity Index (CDAI) Clinical Response by Visit
Description: The Crohn's Disease Activity Index (CDAI) is a composite instrument that includes participant symptoms evaluated over 7 days (abdominal pain, stool frequency and general well-being), as well as physical and laboratory findings. These items are scored individually, weighted, and do not contribute equally to the overall score. The CDAI is derived from summing up the weighted individual scores of eight items. CDAI approximately ranges from 0 to 600 with higher scores indicating more severe disease. Clinical response is defined as CDAI score < 150 or a reduction from baseline of at least 100 points. Baseline is defined as the last measurement prior to the first dose of the study drug in the feeder study NCT02031276 (Boehringer Ingelheim trial 1311.6/AbbVie M15-993).
Time Frame: Weeks 0, 4, 8, 16, 24, 32, 40, 48, 56, 64, 72, 80, 88, 96, 104, 112, 120, 128, 136, 144, 152, 160, 168, 176, and 184
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Risankizumab 600 mg IV | Risankizumab 180 mg SC
Number analyzed (Participants) | 4 | 65
percentage of participants
  Week 0 | 50.00 | 90.77
  Week 4: number analyzed (Participants) | 4 | 0
  Week 4 | 75.00 |
  Week 8 | 100.00 | 98.46
  Week 16: number analyzed (Participants) | 0 | 64
  Week 16 |  | 92.19
  Week 24: number analyzed (Participants) | 0 | 63
  Week 24 |  | 95.24
  Week 32: number analyzed (Participants) | 0 | 61
  Week 32 |  | 95.08
  Week 40: number analyzed (Participants) | 0 | 60
  Week 40 |  | 96.67
  Week 48: number analyzed (Participants) | 0 | 58
  Week 48 |  | 94.83
  Week 56: number analyzed (Participants) | 0 | 57
  Week 56 |  | 92.98
  Week 64: number analyzed (Participants) | 0 | 55
  Week 64 |  | 96.36
  Week 72: number analyzed (Participants) | 0 | 54
  Week 72 |  | 94.44
  Week 80: number analyzed (Participants) | 0 | 53
  Week 80 |  | 92.45
  Week 88: number analyzed (Participants) | 0 | 51
  Week 88 |  | 92.16
  Week 96: number analyzed (Participants) | 0 | 52
  Week 96 |  | 92.31
  Week 104: number analyzed (Participants) | 0 | 49
  Week 104 |  | 93.88
  Week 112: number analyzed (Participants) | 0 | 48
  Week 112 |  | 93.75
  Week 120: number analyzed (Participants) | 0 | 48
  Week 120 |  | 93.75
  Week 128: number analyzed (Participants) | 0 | 46
  Week 128 |  | 93.48
  Week 136: number analyzed (Participants) | 0 | 39
  Week 136 |  | 92.31
  Week 144: number analyzed (Participants) | 0 | 37
  Week 144 |  | 91.89
  Week 152: number analyzed (Participants) | 0 | 30
  Week 152 |  | 93.33
  Week 160: number analyzed (Participants) | 0 | 23
  Week 160 |  | 91.30
  Week 168: number analyzed (Participants) | 0 | 17
  Week 168 |  | 82.35
  Week 176: number analyzed (Participants) | 0 | 10
  Week 176 |  | 80.00
  Week 184: number analyzed (Participants) | 0 | 5
  Week 184 |  | 80.00

4. Secondary Outcome: Percentage of Participants Achieving Patient Reported Outcome 2 (PRO-2) Remission by Visit
Description: The PRO-2 is calculated based on the sum of the weighted patient-reported subscores of CDAI for liquid or soft stool frequency [SF] plus abdominal pain [AP] in the 7 days prior to the study visit. The PRO-2 score is calculated by adding the values of the summed stool frequency scores multiplied by 2 plus the summed abdominal pain scores multiplied by 5. The SF and AP score at an assessment visit was the average of the daily values reported during the 7 days preceding the scheduled assessment visit. PRO-2 scores range from 0 to no upper limit with higher scores indicating more severe disease. Remission is defined as PRO-2 score < 75.
Time Frame: Weeks 0, 4, 8, 16, 24, 32, 40, 48, 56, 64, 72, 80, 88, 96, 104, 112, 120, 128, 136, 144, 152, 160, 168, 176, and 184
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Risankizumab 600 mg IV | Risankizumab 180 mg SC
Number analyzed (Participants) | 4 | 65
percentage of participants
  Week 0 | 25.00 | 73.85
  Week 4: number analyzed (Participants) | 4 | 0
  Week 4 | 25.00 |
  Week 8 | 50.00 | 80.00
  Week 16: number analyzed (Participants) | 0 | 64
  Week 16 |  | 78.13
  Week 24: number analyzed (Participants) | 0 | 63
  Week 24 |  | 77.78
  Week 32: number analyzed (Participants) | 0 | 61
  Week 32 |  | 85.25
  Week 40: number analyzed (Participants) | 0 | 60
  Week 40 |  | 83.33
  Week 48: number analyzed (Participants) | 0 | 58
  Week 48 |  | 82.76
  Week 56: number analyzed (Participants) | 0 | 57
  Week 56 |  | 87.72
  Week 64: number analyzed (Participants) | 0 | 55
  Week 64 |  | 81.82
  Week 72: number analyzed (Participants) | 0 | 54
  Week 72 |  | 81.48
  Week 80: number analyzed (Participants) | 0 | 53
  Week 80 |  | 81.13
  Week 88: number analyzed (Participants) | 0 | 51
  Week 88 |  | 82.35
  Week 96: number analyzed (Participants) | 0 | 52
  Week 96 |  | 84.62
  Week 104: number analyzed (Participants) | 0 | 49
  Week 104 |  | 85.71
  Week 112: number analyzed (Participants) | 0 | 48
  Week 112 |  | 91.67
  Week 120: number analyzed (Participants) | 0 | 48
  Week 120 |  | 85.42
  Week 128: number analyzed (Participants) | 0 | 46
  Week 128 |  | 89.13
  Week 136: number analyzed (Participants) | 0 | 40
  Week 136 |  | 87.50
  Week 144: number analyzed (Participants) | 0 | 37
  Week 144 |  | 86.49
  Week 152: number analyzed (Participants) | 0 | 30
  Week 152 |  | 86.67
  Week 160: number analyzed (Participants) | 0 | 23
  Week 160 |  | 73.91
  Week 168: number analyzed (Participants) | 0 | 18
  Week 168 |  | 77.78
  Week 176: number analyzed (Participants) | 0 | 10
  Week 176 |  | 60.00
  Week 184: number analyzed (Participants) | 0 | 5
  Week 184 |  | 40.00

5. Secondary Outcome: Percentage of Participants Achieving Patient Reported Outcome 2 (PRO-2) Response by Visit
Description: The PRO-2 is calculated based on the sum of the weighted patient-reported subscores of CDAI for liquid or soft stool frequency [SF] plus abdominal pain [AP] in the 7 days prior to the study visit. The PRO-2 score is calculated by adding the values of the summed stool frequency scores multiplied by 2 plus the summed abdominal pain scores multiplied by 5. The SF and AP score at an assessment visit was the average of the daily values reported during the 7 days preceding the scheduled assessment visit. PRO-2 scores range from 0 to no upper limit with higher scores indicating more severe disease. PRO-2 response is defined as a decrease from baseline of 50 points or more. Baseline is defined as the last measurement prior to the first dose of the study drug in the feeder study NCT02031276 (Boehringer Ingelheim trial 1311.6/AbbVie M15-993).
Time Frame: Weeks 0, 4, 8, 16, 24, 32, 40, 48, 56, 64, 72, 80, 88, 96, 104, 112, 120, 128, 136, 144, 152, 160, 168, 176, and 184
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Risankizumab 600 mg IV | Risankizumab 180 mg SC
Number analyzed (Participants) | 4 | 65
percentage of participants
  Week 0 | 50.00 | 83.08
  Week 4: number analyzed (Participants) | 4 | 0
  Week 4 | 50.00 |
  Week 8 | 50.00 | 86.15
  Week 16: number analyzed (Participants) | 0 | 64
  Week 16 |  | 90.63
  Week 24: number analyzed (Participants) | 0 | 63
  Week 24 |  | 92.06
  Week 32: number analyzed (Participants) | 0 | 61
  Week 32 |  | 86.89
  Week 40: number analyzed (Participants) | 0 | 60
  Week 40 |  | 98.33
  Week 48: number analyzed (Participants) | 0 | 58
  Week 48 |  | 93.10
  Week 56: number analyzed (Participants) | 0 | 57
  Week 56 |  | 91.23
  Week 64: number analyzed (Participants) | 0 | 55
  Week 64 |  | 90.91
  Week 72: number analyzed (Participants) | 0 | 54
  Week 72 |  | 88.89
  Week 80: number analyzed (Participants) | 0 | 53
  Week 80 |  | 88.68
  Week 88: number analyzed (Participants) | 0 | 51
  Week 88 |  | 86.27
  Week 96: number analyzed (Participants) | 0 | 52
  Week 96 |  | 88.46
  Week 104: number analyzed (Participants) | 0 | 49
  Week 104 |  | 87.76
  Week 112: number analyzed (Participants) | 0 | 48
  Week 112 |  | 87.50
  Week 120: number analyzed (Participants) | 0 | 48
  Week 120 |  | 91.67
  Week 128: number analyzed (Participants) | 0 | 46
  Week 128 |  | 91.30
  Week 136: number analyzed (Participants) | 0 | 40
  Week 136 |  | 92.50
  Week 144: number analyzed (Participants) | 0 | 37
  Week 144 |  | 89.19
  Week 152: number analyzed (Participants) | 0 | 30
  Week 152 |  | 93.33
  Week 160: number analyzed (Participants) | 0 | 23
  Week 160 |  | 86.96
  Week 168: number analyzed (Participants) | 0 | 18
  Week 168 |  | 83.33
  Week 176: number analyzed (Participants) | 0 | 10
  Week 176 |  | 100.00
  Week 184: number analyzed (Participants) | 0 | 5
  Week 184 |  | 100.00

6. Secondary Outcome: Percentage of Participants Achieving Crohn's Disease Endoscopic Index of Severity (CDEIS) Remission by Visit
Description: CDEIS is an index for determining the severity of Crohn's disease. The CDEIS considers deep ulcerations, superficial ulcerations, ulcerated and non-ulcerated surface, and the presence of ulcerated/non-ulcerated stenosis evaluated in 5 pre-defined segments of the colon (ileum, ascending colon, transverse colon, descending colon and sigmoid loop, and rectum). The score ranges from 0 to 44 where higher scores indicate more severe endoscopic activity. Remission is defined as a score of 4 or less, by visit (or for participants with initial isolated ileitis a score of 2 or less).
Time Frame: Weeks 0, 48, 104, 152, and 200
Population: Observed case (OC) analysis was performed on the intent-to-treat (ITT) SC analysis set, which consisted of all participants who received at least one dose of risankizumab SC in the current study.
Measure: Number; unit: percentage of participants
Arm/Group | Risankizumab 180 mg SC
Number analyzed (Participants) | 63
percentage of participants
  Week 0 | 42.86
  Week 48: number analyzed (Participants) | 62
  Week 48 | 56.45
  Week 104: number analyzed (Participants) | 43
  Week 104 | 62.79
  Week 152: number analyzed (Participants) | 39
  Week 152 | 58.97
  Week 200: number analyzed (Participants) | 7
  Week 200 | 85.71

7. Secondary Outcome: Percentage of Participants Achieving Crohn's Disease Endoscopic Index of Severity (CDEIS) Response by Visit
Description: CDEIS is an index for determining the severity of Crohn's disease. The CDEIS considers deep ulcerations, superficial ulcerations, ulcerated and non-ulcerated surface, and the presence of ulcerated/non-ulcerated stenosis evaluated in 5 pre-defined segments of the colon (ileum, ascending colon, transverse colon, descending colon and sigmoid loop, and rectum). The score ranges from 0 to 44 where higher scores indicate more severe endoscopic activity. Response is defined as a score of 7 or less (or for participants with initial isolated ileitis > 50% reduction from baseline). Baseline is defined as the last measurement prior to the first dose of the study drug in the feeder study NCT02031276 (Boehringer Ingelheim trial 1311.6/AbbVie M15-993).
Time Frame: Weeks 0, 48, 104, 152, and 200
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | Risankizumab 180 mg SC
Number analyzed (Participants) | 63
percentage of participants
  Week 0 | 58.73
  Week 48: number analyzed (Participants) | 62
  Week 48 | 72.58
  Week 104: number analyzed (Participants) | 43
  Week 104 | 81.40
  Week 152: number analyzed (Participants) | 39
  Week 152 | 82.05
  Week 200: number analyzed (Participants) | 7
  Week 200 | 100.00

8. Secondary Outcome: Percentage of Participants With Mucosal Healing by Visit
Description: Mucosal healing is defined as Crohn's Disease Endoscopy Index of Severity (CDEIS) ulcerations sub-score (deep ulceration, superficial ulceration, ulcerated stenosis) of 0 as evaluated in 5 pre-defined segments of the colon (ileum, ascending colon, transverse colon, descending colon and sigmoid loop, and rectum). The overall CDEIS score ranges from 0 to 44 where higher scores indicate more severe endoscopic activity.
Time Frame: Weeks 0, 48, 104, 152, and 200
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | Risankizumab 180 mg SC
Number analyzed (Participants) | 64
percentage of participants
  Week 0 | 29.69
  Week 48: number analyzed (Participants) | 62
  Week 48 | 35.48
  Week 104: number analyzed (Participants) | 43
  Week 104 | 39.53
  Week 152: number analyzed (Participants) | 39
  Week 152 | 43.59
  Week 200: number analyzed (Participants) | 7
  Week 200 | 42.86

9. Secondary Outcome: Percentage of Participants Achieving Deep Remission by Visit
Description: Deep remission is defined as clinical remission (CDAI < 150) and CDEIS remission (CDEIS score of 4 or less, by visit or for participants with initial isolated ileitis a score of 2 or less).
Time Frame: Weeks 0, 48, 104, 152, and 200
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | Risankizumab 180 mg SC
Number analyzed (Participants) | 63
percentage of participants
  Week 0 | 34.92
  Week 48: number analyzed (Participants) | 61
  Week 48 | 47.54
  Week 104: number analyzed (Participants) | 43
  Week 104 | 53.49
  Week 152: number analyzed (Participants) | 35
  Week 152 | 42.86
  Week 200: number analyzed (Participants) | 1
  Week 200 | 0.00

10. Secondary Outcome: Percentage of Participants Achieving Inflammatory Bowel Disease Questionnaire (IBDQ) Remission by Visit
Description: The Inflammatory Bowel Disease Questionnaire (IBDQ) measures the effects of inflammatory bowel disease on daily function and quality of life. The IBDQ consists of 32 questions which address symptoms as a result of Crohn's disease: bowel symptoms (loose stools, abdominal pain), systemic symptoms (fatigue, altered sleep pattern), social function (work attendance, need to cancel social events), and emotional function (anger, depression, irritability). Each question is answered on a scale from 1 (all the time) to 7 (none of the time); the total score ranges from 32 (worst) to 224 (best). IBDQ remission is defined as IBDQ total score > 170 points.
Time Frame: Weeks 0, 24, 48, 72, 96, 120, 144, 168, and 192
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | Risankizumab 180 mg SC
Number analyzed (Participants) | 65
percentage of participants
  Week 0: number analyzed (Participants) | 64
  Week 0 | 62.50
  Week 24 | 58.46
  Week 48: number analyzed (Participants) | 60
  Week 48 | 70.00
  Week 72: number analyzed (Participants) | 52
  Week 72 | 69.23
  Week 96: number analyzed (Participants) | 51
  Week 96 | 72.55
  Week 120: number analyzed (Participants) | 48
  Week 120 | 70.83
  Week 144: number analyzed (Participants) | 40
  Week 144 | 65.00
  Week 168: number analyzed (Participants) | 23
  Week 168 | 69.57
  Week 192: number analyzed (Participants) | 6
  Week 192 | 66.67

11. Secondary Outcome: Percentage of Participants Achieving Inflammatory Bowel Disease Questionnaire (IBDQ) Response by Visit
Description: The Inflammatory Bowel Disease Questionnaire (IBDQ) measures the effects of inflammatory bowel disease on daily function and quality of life. The IBDQ consists of 32 questions which address symptoms as a result of Crohn's disease: bowel symptoms (loose stools, abdominal pain), systemic symptoms (fatigue, altered sleep pattern), social function (work attendance, need to cancel social events), and emotional function (anger, depression, irritability). Each question is answered on a scale from 1 (all the time) to 7 (none of the time); the total score ranges from 32 (worst) to 224 (best). IBDQ response is defined as increase in IBDQ total score >16 points from baseline. Baseline is defined as the last measurement prior to the first dose of the study drug in the feeder study NCT02031276 (Boehringer Ingelheim trial 1311.6/AbbVie M15-993).
Time Frame: Weeks 0, 24, 48, 72, 96, 120, 144, 168, and 192
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | Risankizumab 180 mg SC
Number analyzed (Participants) | 65
percentage of participants
  Week 0: number analyzed (Participants) | 64
  Week 0 | 92.19
  Week 24 | 89.23
  Week 48: number analyzed (Participants) | 60
  Week 48 | 95.00
  Week 72: number analyzed (Participants) | 52
  Week 72 | 88.46
  Week 96: number analyzed (Participants) | 51
  Week 96 | 90.20
  Week 120: number analyzed (Participants) | 48
  Week 120 | 95.83
  Week 144: number analyzed (Participants) | 40
  Week 144 | 92.50
  Week 168: number analyzed (Participants) | 23
  Week 168 | 86.96
  Week 192: number analyzed (Participants) | 6
  Week 192 | 100.00

12. Secondary Outcome: Mean Change From Baseline in Crohn's Disease Activity Index (CDAI) by Visit
Description: The Crohn's Disease Activity Index (CDAI) is a composite instrument that includes participant symptoms evaluated over 7 days (abdominal pain, stool frequency and general well-being), as well as physical and laboratory findings. These items are scored individually, weighted, and do not contribute equally to the overall score. The CDAI is derived from summing up the weighted individual scores of eight items. CDAI approximately ranges from 0 to 600 with higher scores indicating more severe disease. Baseline is defined as the last measurement prior to the first dose of the study drug in the feeder study NCT02031276 (Boehringer Ingelheim trial 1311.6/AbbVie M15-993). A negative change from baseline indicates improvement.
Time Frame: Weeks 0, 4, 8, 16, 24, 32, 40, 48, 56, 64, 72, 80, 88, 96, 104, 112, 120, 128, 136, 144, 152, 160, 168, 176, and 184
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Risankizumab 600 mg IV | Risankizumab 180 mg SC
Number analyzed (Participants) | 4 | 65
units on a scale
  Week 0 | -50.70 (84.565) | -198.47 (101.762)
  Week 4: number analyzed (Participants) | 4 | 0
  Week 4 | -92.68 (40.688) |
  Week 8 | -119.40 (32.967) | -206.75 (83.580)
  Week 16: number analyzed (Participants) | 0 | 64
  Week 16 |  | -205.93 (92.837)
  Week 24: number analyzed (Participants) | 0 | 63
  Week 24 |  | -194.34 (82.840)

13. Secondary Outcome: Mean Change From Baseline in Patient Reported Outcome 2 (PRO-2) Scores by Visit
Description: The PRO-2 is calculated based on the sum of the weighted patient-reported subscores of CDAI for liquid or soft stool frequency [SF] plus abdominal pain [AP] in the 7 days prior to the study visit. The PRO-2 score is calculated by adding the values of the summed stool frequency scores multiplied by 2 plus the summed abdominal pain scores multiplied by 5. The SF and AP score at an assessment visit was the average of the daily values reported during the 7 days preceding the scheduled assessment visit. PRO-2 scores range from 0 to no upper limit with higher scores indicating more severe disease. Baseline is defined as the last measurement prior to the first dose of the study drug in the feeder study NCT02031276 (Boehringer Ingelheim trial 1311.6/AbbVie M15-993). A negative change from baseline indicates improvement.
Time Frame: Weeks 0, 4, 8, 16, 24, 32, 40, 48, 56, 64, 72, 80, 88, 96, 104, 112, 120, 128, 136, 144, 152, 160, 168, 176, and 184
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Risankizumab 600 mg IV | Risankizumab 180 mg SC
Number analyzed (Participants) | 4 | 65
units on a scale
  Week 0 | -27.75 (48.979) | -105.46 (58.807)
  Week 4: number analyzed (Participants) | 4 | 0
  Week 4 | -35.25 (27.011) |
  Week 8 | -53.75 (24.405) | -109.53 (49.419)
  Week 16: number analyzed (Participants) | 0 | 64
  Week 16 |  | -108.32 (52.848)
  Week 24: number analyzed (Participants) | 0 | 63
  Week 24 |  | -105.40 (50.167)
  Week 32: number analyzed (Participants) | 0 | 61
  Week 32 |  | -109.41 (56.459)
  Week 40: number analyzed (Participants) | 0 | 60
  Week 40 |  | -116.33 (43.511)
  Week 48: number analyzed (Participants) | 0 | 58
  Week 48 |  | -111.29 (48.048)
  Week 56: number analyzed (Participants) | 0 | 57
  Week 56 |  | -115.54 (51.279)
  Week 64: number analyzed (Participants) | 0 | 55
  Week 64 |  | -113.02 (57.338)
  Week 72: number analyzed (Participants) | 0 | 54
  Week 72 |  | -112.11 (56.819)
  Week 80: number analyzed (Participants) | 0 | 53
  Week 80 |  | -106.42 (58.710)
  Week 88: number analyzed (Participants) | 0 | 51
  Week 88 |  | -108.67 (51.214)
  Week 96: number analyzed (Participants) | 0 | 52
  Week 96 |  | -109.81 (50.927)
  Week 104: number analyzed (Participants) | 0 | 49
  Week 104 |  | -109.10 (49.562)
  Week 112: number analyzed (Participants) | 0 | 48
  Week 112 |  | -109.75 (52.951)
  Week 120: number analyzed (Participants) | 0 | 48
  Week 120 |  | -111.10 (47.360)
  Week 128: number analyzed (Participants) | 0 | 46
  Week 128 |  | -113.02 (50.738)
  Week 136: number analyzed (Participants) | 0 | 40
  Week 136 |  | -113.00 (51.575)
  Week 144: number analyzed (Participants) | 0 | 37
  Week 144 |  | -115.35 (53.460)
  Week 152: number analyzed (Participants) | 0 | 30
  Week 152 |  | -109.17 (56.659)
  Week 160: number analyzed (Participants) | 0 | 23
  Week 160 |  | -96.70 (54.018)
  Week 168: number analyzed (Participants) | 0 | 18
  Week 168 |  | -111.09 (55.287)
  Week 176: number analyzed (Participants) | 0 | 10
  Week 176 |  | -103.06 (42.717)
  Week 184: number analyzed (Participants) | 0 | 5
  Week 184 |  | -129.13 (70.484)

14. Secondary Outcome: Mean Change From Baseline in Crohn's Disease Endoscopic Index of Severity (CDEIS) by Visit
Description: CDEIS is an index for determining the severity of Crohn's disease. The CDEIS considers deep ulcerations, superficial ulcerations, ulcerated and non-ulcerated surface, and the presence of ulcerated/non-ulcerated stenosis evaluated in 5 pre-defined segments of the colon (ileum, ascending colon, transverse colon, descending colon and sigmoid loop, and rectum). The score ranges from 0 to 44 where higher scores indicate more severe endoscopic activity. Baseline is defined as the last measurement prior to the first dose of the study drug in the feeder study NCT02031276 (Boehringer Ingelheim trial 1311.6/AbbVie M15-993). A negative change from baseline indicates improvement.
Time Frame: Weeks 0, 48, 104, 152, and 200
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Risankizumab 180 mg SC
Number analyzed (Participants) | 63
units on a scale
  Week 0 | -8.08 (5.973)
  Week 48: number analyzed (Participants) | 62
  Week 48 | -9.32 (6.014)
  Week 104: number analyzed (Participants) | 43
  Week 104 | -9.24 (6.035)
  Week 152: number analyzed (Participants) | 39
  Week 152 | -9.75 (7.254)
  Week 200: number analyzed (Participants) | 7
  Week 200 | -10.76 (5.209)

15. Secondary Outcome: Mean Change From Baseline in Simple Endoscopic Score (SES-CD) by Visit
Description: SES-CD is calculated based the sum of individual segment values for four endoscopic variables (presence and size of ulcers, ulcerated surface, affected surface and presence of narrowing). Each variable in each segment is scored 0 to 3 resulting in SES-CD values ranging from 0 to 56 with higher scores indicating more severe disease. Baseline is defined as the last measurement prior to the first dose of the study drug in the feeder study NCT02031276 (Boehringer Ingelheim trial 1311.6/AbbVie M15-993). A negative change from baseline indicates improvement.
Time Frame: Weeks 0, 48, 104, 152, and 200
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Risankizumab 180 mg SC
Number analyzed (Participants) | 63
units on a scale
  Week 0 | -9.63 (8.001)
  Week 48: number analyzed (Participants) | 62
  Week 48 | -12.35 (7.753)
  Week 104: number analyzed (Participants) | 43
  Week 104 | -11.56 (8.060)
  Week 152: number analyzed (Participants) | 39
  Week 152 | -12.63 (9.139)
  Week 200: number analyzed (Participants) | 7
  Week 200 | -13.36 (7.521)

16. Secondary Outcome: Mean Change From Baseline in Stool Frequency (SF) By Visit
Description: Participants were asked to record the frequency of liquid stools on a daily basis. The number of liquid stools in the prior 7 days was summed. Baseline is defined as the last measurement prior to the first dose of the study drug in the feeder study NCT02031276 (Boehringer Ingelheim trial 1311.6/AbbVie M15-993). Negative values indicate improvement from baseline.
Time Frame: Weeks 0, 4, 8, 16, 24, 32, 40, 48, 56, 64, 72, 80, 88, 96, 104, 112, 120, 128, 136, 144, 152, 160, 168, 176, and 184
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: number of liquid stools in prior 7 days
Arm/Group | Risankizumab 600 mg IV | Risankizumab 180 mg SC
Number analyzed (Participants) | 4 | 65
number of liquid stools in prior 7 days
  Week 0 | -0.46 (2.319) | -4.13 (3.273)
  Week 4: number analyzed (Participants) | 4 | 0
  Week 4 | -0.46 (1.584) |
  Week 8 | -1.07 (1.421) | -4.22 (3.160)
  Week 16: number analyzed (Participants) | 0 | 64
  Week 16 |  | -4.10 (3.223)
  Week 24: number analyzed (Participants) | 0 | 63
  Week 24 |  | -4.19 (3.209)
  Week 32: number analyzed (Participants) | 0 | 61
  Week 32 |  | -4.08 (3.536)
  Week 40: number analyzed (Participants) | 0 | 60
  Week 40 |  | -4.58 (3.037)
  Week 48: number analyzed (Participants) | 0 | 58
  Week 48 |  | -4.31 (3.278)
  Week 56: number analyzed (Participants) | 0 | 57
  Week 56 |  | -4.48 (3.282)
  Week 64: number analyzed (Participants) | 0 | 55
  Week 64 |  | -4.41 (3.514)
  Week 72: number analyzed (Participants) | 0 | 54
  Week 72 |  | -4.25 (3.513)
  Week 80: number analyzed (Participants) | 0 | 53
  Week 80 |  | -4.00 (3.469)
  Week 88: number analyzed (Participants) | 0 | 51
  Week 88 |  | -4.04 (3.331)
  Week 96: number analyzed (Participants) | 0 | 52
  Week 96 |  | -4.27 (3.037)
  Week 104: number analyzed (Participants) | 0 | 49
  Week 104 |  | -4.00 (2.943)
  Week 112: number analyzed (Participants) | 0 | 48
  Week 112 |  | -3.91 (2.951)
  Week 120: number analyzed (Participants) | 0 | 48
  Week 120 |  | -3.99 (2.840)
  Week 128: number analyzed (Participants) | 0 | 46
  Week 128 |  | -4.05 (3.060)
  Week 136: number analyzed (Participants) | 0 | 40
  Week 136 |  | -3.95 (3.137)
  Week 144: number analyzed (Participants) | 0 | 37
  Week 144 |  | -4.13 (3.308)
  Week 152: number analyzed (Participants) | 0 | 30
  Week 152 |  | -4.00 (3.150)
  Week 160: number analyzed (Participants) | 0 | 23
  Week 160 |  | -3.71 (3.044)
  Week 168: number analyzed (Participants) | 0 | 18
  Week 168 |  | -4.08 (3.353)
  Week 176: number analyzed (Participants) | 0 | 10
  Week 176 |  | -3.61 (2.583)
  Week 184: number analyzed (Participants) | 0 | 5
  Week 184 |  | -4.50 (3.881)

17. Secondary Outcome: Mean Change From Baseline in Abdominal Pain (AP) Score By Visit
Description: Participants were asked to rate and record daily abdominal pain on a scale of 0 to 3 [none (0), mild (1), moderate (2) and severe (3)]. The ratings in the prior 7 days were summed. Baseline is defined as the last measurement prior to the first dose of the study drug in the feeder study NCT02031276 (Boehringer Ingelheim trial 1311.6/AbbVie M15-993). Negative values indicate improvement from baseline.
Time Frame: Weeks 0, 4, 8, 16, 24, 32, 40, 48, 56, 64, 72, 80, 88, 96, 104, 112, 120, 128, 136, 144, 152, 160, 168, 176, and 184
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Risankizumab 600 mg IV | Risankizumab 180 mg SC
Number analyzed (Participants) | 4 | 65
units on a scale
  Week 0 | -0.61 (1.006) | -1.36 (0.885)
  Week 4: number analyzed (Participants) | 4 | 0
  Week 4 | -0.82 (0.768) |
  Week 8 | -1.11 (0.357) | -1.44 (0.746)
  Week 16: number analyzed (Participants) | 0 | 64
  Week 16 |  | -1.45 (0.773)
  Week 24: number analyzed (Participants) | 0 | 63
  Week 24 |  | -1.33 (0.804)
  Week 32: number analyzed (Participants) | 0 | 61
  Week 32 |  | -1.49 (0.760)
  Week 40: number analyzed (Participants) | 0 | 60
  Week 40 |  | -1.49 (0.766)
  Week 48: number analyzed (Participants) | 0 | 58
  Week 48 |  | -1.46 (0.720)
  Week 56: number analyzed (Participants) | 0 | 57
  Week 56 |  | -1.51 (0.815)
  Week 64: number analyzed (Participants) | 0 | 55
  Week 64 |  | -1.47 (0.825)
  Week 72: number analyzed (Participants) | 0 | 54
  Week 72 |  | -1.50 (0.839)
  Week 80: number analyzed (Participants) | 0 | 53
  Week 80 |  | -1.44 (0.816)
  Week 88: number analyzed (Participants) | 0 | 51
  Week 88 |  | -1.49 (0.787)
  Week 96: number analyzed (Participants) | 0 | 52
  Week 96 |  | -1.43 (0.881)
  Week 104: number analyzed (Participants) | 0 | 49
  Week 104 |  | -1.52 (0.861)
  Week 112: number analyzed (Participants) | 0 | 48
  Week 112 |  | -1.57 (0.890)
  Week 120: number analyzed (Participants) | 0 | 48
  Week 120 |  | -1.58 (0.735)
  Week 128: number analyzed (Participants) | 0 | 46
  Week 128 |  | -1.61 (0.776)
  Week 136: number analyzed (Participants) | 0 | 40
  Week 136 |  | -1.65 (0.792)
  Week 144: number analyzed (Participants) | 0 | 37
  Week 144 |  | -1.64 (0.836)
  Week 152: number analyzed (Participants) | 0 | 30
  Week 152 |  | -1.52 (0.833)
  Week 160: number analyzed (Participants) | 0 | 23
  Week 160 |  | -1.28 (0.788)
  Week 168: number analyzed (Participants) | 0 | 18
  Week 168 |  | -1.54 (0.657)
  Week 176: number analyzed (Participants) | 0 | 10
  Week 176 |  | -1.50 (0.670)
  Week 184: number analyzed (Participants) | 0 | 5
  Week 184 |  | -1.89 (0.921)

18. Secondary Outcome: Mean Change From Baseline in Inflammatory Bowel Disease Questionnaire (IBDQ) Total Score by Visit
Description: The Inflammatory Bowel Disease Questionnaire (IBDQ) measures the effects of inflammatory bowel disease on daily function and quality of life. The IBDQ consists of 32 questions which address symptoms as a result of Crohn's disease: bowel symptoms (loose stools, abdominal pain), systemic symptoms (fatigue, altered sleep pattern), social function (work attendance, need to cancel social events), and emotional function (anger, depression, irritability). Each question is answered on a scale from 1 (all the time) to 7 (none of the time); the total score ranges from 32 (worst) to 224 (best). Baseline is defined as the last measurement prior to the first dose of the study drug in the feeder study NCT02031276 (Boehringer Ingelheim trial 1311.6/AbbVie M15-993). Positive values indicate improvement from baseline.
Time Frame: Weeks 0, 24, 48, 72, 96, 120, 144, 168, and 192
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Risankizumab 180 mg SC
Number analyzed (Participants) | 65
units on a scale
  Week 0: number analyzed (Participants) | 64
  Week 0 | 62.48 (38.791)
  Week 24 | 58.72 (35.626)
  Week 48: number analyzed (Participants) | 60
  Week 48 | 64.03 (33.039)
  Week 72: number analyzed (Participants) | 52
  Week 72 | 64.14 (42.229)
  Week 96: number analyzed (Participants) | 51
  Week 96 | 62.38 (39.220)
  Week 120: number analyzed (Participants) | 48
  Week 120 | 67.28 (34.390)
  Week 144: number analyzed (Participants) | 40
  Week 144 | 61.34 (34.894)
  Week 168: number analyzed (Participants) | 23
  Week 168 | 56.36 (33.035)
  Week 192: number analyzed (Participants) | 6
  Week 192 | 71.17 (41.911)

19. Secondary Outcome: Mean Change From Baseline in Inflammatory Bowel Disease Questionnaire (IBDQ) Bowel Symptom Domain Score by Visit
Description: as for outcome 18
Time Frame: Weeks 0, 24, 48, 72, 96, 120, 144, 168, and 192
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Risankizumab 180 mg SC
Number analyzed (Participants) | 65
units on a scale
  Week 0: number analyzed (Participants) | 64
  Week 0 | 20.44 (11.680)
  Week 24 | 18.26 (11.587)
  Week 48: number analyzed (Participants) | 60
  Week 48 | 20.29 (10.861)
  Week 72: number analyzed (Participants) | 52
  Week 72 | 20.64 (12.547)
  Week 96: number analyzed (Participants) | 51
  Week 96 | 19.12 (13.064)
  Week 120: number analyzed (Participants) | 48
  Week 120 | 22.25 (10.473)
  Week 144: number analyzed (Participants) | 40
  Week 144 | 20.46 (10.639)
  Week 168: number analyzed (Participants) | 23
  Week 168 | 18.44 (10.658)
  Week 192: number analyzed (Participants) | 6
  Week 192 | 22.67 (14.962)

20. Secondary Outcome: Mean Change From Baseline in Inflammatory Bowel Disease Questionnaire (IBDQ) Systemic System Domain Score by Visit
Description: as for outcome 18
Time Frame: Weeks 0, 24, 48, 72, 96, 120, 144, 168, and 192
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Risankizumab 180 mg SC
Number analyzed (Participants) | 65
units on a scale
  Week 0: number analyzed (Participants) | 64
  Week 0 | 9.9 (6.66)
  Week 24 | 9.1 (6.44)
  Week 48: number analyzed (Participants) | 60
  Week 48 | 9.6 (6.08)
  Week 72: number analyzed (Participants) | 52
  Week 72 | 10.1 (7.36)
  Week 96: number analyzed (Participants) | 51
  Week 96 | 10.3 (5.80)
  Week 120: number analyzed (Participants) | 48
  Week 120 | 9.8 (6.16)
  Week 144: number analyzed (Participants) | 40
  Week 144 | 8.9 (6.02)
  Week 168: number analyzed (Participants) | 23
  Week 168 | 8.2 (5.10)
  Week 192: number analyzed (Participants) | 6
  Week 192 | 11.8 (4.62)

21. Secondary Outcome: Mean Change From Baseline in Inflammatory Bowel Disease Questionnaire (IBDQ) Social Function Domain Score by Visit
Description: as for outcome 18
Time Frame: Weeks 0, 24, 48, 72, 96, 120, 144, 168, and 192
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Risankizumab 180 mg SC
Number analyzed (Participants) | 65
units on a scale
  Week 0: number analyzed (Participants) | 64
  Week 0 | 11.04 (8.230)
  Week 24 | 10.57 (7.652)
  Week 48: number analyzed (Participants) | 60
  Week 48 | 11.64 (7.487)
  Week 72: number analyzed (Participants) | 52
  Week 72 | 11.20 (8.731)
  Week 96: number analyzed (Participants) | 51
  Week 96 | 10.59 (8.556)
  Week 120: number analyzed (Participants) | 48
  Week 120 | 11.92 (7.347)
  Week 144: number analyzed (Participants) | 40
  Week 144 | 10.93 (8.309)
  Week 168: number analyzed (Participants) | 23
  Week 168 | 10.87 (9.503)
  Week 192: number analyzed (Participants) | 6
  Week 192 | 11.67 (9.266)

22. Secondary Outcome: Mean Change From Baseline in Inflammatory Bowel Disease Questionnaire (IBDQ) Emotional Function Domain Score by Visit
Description: as for outcome 18
Time Frame: Weeks 0, 24, 48, 72, 96, 120, 144, 168, and 192
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Risankizumab 180 mg SC
Number analyzed (Participants) | 65
units on a scale
  Week 0: number analyzed (Participants) | 64
  Week 0 | 21.09 (16.820)
  Week 24 | 20.79 (15.632)
  Week 48: number analyzed (Participants) | 60
  Week 48 | 22.55 (14.965)
  Week 72: number analyzed (Participants) | 52
  Week 72 | 22.23 (17.912)
  Week 96: number analyzed (Participants) | 51
  Week 96 | 22.41 (17.075)
  Week 120: number analyzed (Participants) | 48
  Week 120 | 23.35 (15.391)
  Week 144: number analyzed (Participants) | 40
  Week 144 | 21.03 (15.044)
  Week 168: number analyzed (Participants) | 23
  Week 168 | 18.87 (14.552)
  Week 192: number analyzed (Participants) | 6
  Week 192 | 25.00 (21.373)

23. Secondary Outcome: Mean Change From Baseline in High-Sensitivity C-reactive Protein (Hs-CRP) by Visit
Description: Concentration of serum high-sensitivity C-reactive Protein (hs-CRP) was analyzed by a central laboratory. It is a general marker of inflammation that is sensitive to acute changes in inflammatory response, and higher levels indicate more inflammation. Baseline is defined as the last measurement prior to the first dose of the study drug in the feeder study NCT02031276 (Boehringer Ingelheim trial 1311.6/AbbVie M15-993). Negative values indicate improvement from baseline.
Time Frame: Weeks 0, 8, 24, 40, 56, 72, 88, 104, 120, 128, 136, 152, 160, 176, and 184
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Risankizumab 180 mg SC
Number analyzed (Participants) | 65
mg/L
  Week 0 | -14.64 (22.842)
  Week 8: number analyzed (Participants) | 64
  Week 8 | -15.84 (22.548)
  Week 24: number analyzed (Participants) | 64
  Week 24 | -12.76 (24.457)
  Week 40: number analyzed (Participants) | 60
  Week 40 | -14.32 (24.080)
  Week 56: number analyzed (Participants) | 57
  Week 56 | -16.11 (24.194)
  Week 72: number analyzed (Participants) | 54
  Week 72 | -14.40 (21.878)
  Week 88: number analyzed (Participants) | 50
  Week 88 | -17.07 (23.312)
  Week 104: number analyzed (Participants) | 50
  Week 104 | -14.44 (20.057)
  Week 120: number analyzed (Participants) | 47
  Week 120 | -13.81 (22.667)
  Week 128: number analyzed (Participants) | 46
  Week 128 | -14.87 (20.133)
  Week 136: number analyzed (Participants) | 40
  Week 136 | -15.78 (20.864)
  Week 152: number analyzed (Participants) | 36
  Week 152 | -17.03 (20.998)
  Week 160: number analyzed (Participants) | 22
  Week 160 | -18.43 (22.147)
  Week 176: number analyzed (Participants) | 15
  Week 176 | -20.49 (25.062)
  Week 184: number analyzed (Participants) | 5
  Week 184 | -25.01 (32.459)

24. Secondary Outcome: Mean Change From Baseline in Fecal Calprotectin (FCP) Profile by Visit
Description: Fecal calprotectin (FCP) is an indicator of inflammation in the colon with higher levels indicative of higher levels of inflammation. Stool samples were analyzed by a central laboratory for fecal calprotectin levels. Baseline is defined as the last measurement prior to the first dose of the study drug in the feeder study NCT02031276 (Boehringer Ingelheim trial 1311.6/AbbVie M15-993). Negative values indicate improvement from baseline.
Time Frame: Weeks 0, 24, 56, 88, 120, 152, and 184
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: μg/g
Arm/Group | Risankizumab 180 mg SC
Number analyzed (Participants) | 65
μg/g
  Week 0 | -1983.9 (3402.12)
  Week 24: number analyzed (Participants) | 57
  Week 24 | -2166.4 (4035.66)
  Week 56: number analyzed (Participants) | 52
  Week 56 | -2277.8 (4104.19)
  Week 88: number analyzed (Participants) | 49
  Week 88 | -2485.9 (4157.37)
  Week 120: number analyzed (Participants) | 40
  Week 120 | -2031.9 (5187.92)
  Week 152: number analyzed (Participants) | 36
  Week 152 | -2631.5 (4589.62)
  Week 184: number analyzed (Participants) | 12
  Week 184 | -4436.1 (7455.55)

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) and serious adverse events (TESAEs) were collected from the first dose of study drug until 140 days after the last dose of study drug in the current study or until the first dose of study drug in NCT03105102 (AbbVie M16-000 Sub-study 3), up to 4 years for participants who rolled-over.
Description: TEAEs and SAEs are defined as any adverse event (AE) with an onset date that is on or after the first dose of study drug until 140 days after the last dose of study drug and were collected whether elicited or spontaneously reported by the participant.
Arm/Group | Risankizumab 600 mg IV | Risankizumab 180 mg SC | All Risankizumab
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/65 | 0/65
Serious Adverse Events (participants affected / at risk) | 0/4 | 23/65 | 23/65
Other Adverse Events (participants affected / at risk) | 2/4 | 52/65 | 52/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Risankizumab 600 mg IV (N=4) | Risankizumab 180 mg SC (N=65) | All Risankizumab (N=65)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (3) | 1 (3)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 1 (1) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Crohn's disease (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2)
Dumping syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Ileal stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Impaired gastric emptying (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Intestinal stenosis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1) | 1 (1)
Anal abscess (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Campylobacter infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 2 (2) | 2 (2)
Peritonitis (Infections and infestations) | 0 (0) | 2 (2) | 2 (2)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Anastomotic leak (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Post procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 2 (2)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Carotid sinus syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Cluster headache (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 1 (1)
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Selective abortion (Surgical and medical procedures) | 0 (0) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Risankizumab 600 mg IV (N=4) | Risankizumab 180 mg SC (N=65) | All Risankizumab (N=65)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 4 (5) | 4 (5)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 12 (13) | 12 (13)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 4 (6) | 5 (7)
Constipation (Gastrointestinal disorders) | 0 (0) | 4 (4) | 4 (4)
Crohn's disease (Gastrointestinal disorders) | 0 (0) | 10 (11) | 10 (11)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 8 (9) | 8 (9)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 4 (4) | 4 (4)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 2 (5) | 2 (6)
Nausea (Gastrointestinal disorders) | 0 (0) | 10 (10) | 10 (10)
Odynophagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 4 (4) | 5 (5)
Fatigue (General disorders) | 0 (0) | 13 (14) | 13 (14)
Ear infection (Infections and infestations) | 0 (0) | 4 (4) | 4 (4)
Gastroenteritis (Infections and infestations) | 0 (0) | 15 (19) | 15 (19)
Influenza (Infections and infestations) | 0 (0) | 8 (11) | 8 (11)
Nasopharyngitis (Infections and infestations) | 1 (2) | 20 (38) | 20 (40)
Oral herpes (Infections and infestations) | 0 (0) | 5 (6) | 5 (6)
Pharyngitis (Infections and infestations) | 0 (0) | 4 (7) | 4 (7)
Rhinitis (Infections and infestations) | 0 (0) | 6 (7) | 6 (7)
Sinusitis (Infections and infestations) | 0 (0) | 5 (6) | 5 (6)
Tooth abscess (Infections and infestations) | 0 (0) | 5 (7) | 5 (7)
Tracheitis (Infections and infestations) | 0 (0) | 4 (5) | 4 (5)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 7 (8) | 7 (9)
Urinary tract infection (Infections and infestations) | 0 (0) | 9 (10) | 9 (10)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 5 (5) | 5 (5)
Alanine aminotransferase increased (Investigations) | 0 (0) | 4 (4) | 4 (4)
Weight increased (Investigations) | 1 (1) | 2 (2) | 2 (3)
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 3 (3)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 4 (4) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 11 (14) | 11 (14)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 8 (10) | 8 (10)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 5 (6) | 5 (6)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 5 (8) | 5 (8)
Headache (Nervous system disorders) | 0 (0) | 9 (15) | 9 (15)
Insomnia (Psychiatric disorders) | 0 (0) | 5 (5) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 6 (10) | 6 (10)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 5 (5) | 5 (5)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (4) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2018-07-25): https://cdn.clinicaltrials.gov/large-docs/59/NCT02513459/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-15): https://cdn.clinicaltrials.gov/large-docs/59/NCT02513459/SAP_001.pdf